CLINICAL TRIAL: NCT02220010
Title: Does a Pancreatic Stent Reduce the Healing Time of Post Operative Pancreatic Fistula (POPF) After Distal Pancreatic Resection - an Open Randomized Clinical Multicenter Trial
Brief Title: Does Post Operative Pancreatic Fistula, After Left Sided Resections, Heal Faster After the Introduction of a Pancreatic Stent?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Lund University Hospital (Other); University Hospital, Linkoeping (Other); Norrlands University Hospital (Other)
Responsible Party: Principal Investigator, John Blomberg, M.D., PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POPF and stenting-002
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Healing Time of Post Operative Pancreatic Fistulas
Keywords: Post operative pancreatic fistulas; Pancreatic stenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pancreatic stent (Experimental): If POPF grade B or C is detected on post operative day 3 or more, a pancreatic stent is endoscopically positioned in the pancreatic duct.
  Interventions: Device: Pancreatic stent
- Drain only (No Intervention): If POPF grade B or C is detected on post operative day 3 or more, only the per-operatively placed drain is used as treatment

INTERVENTIONS:
Device: Pancreatic stent — The plastic stent is introduced in the pancreatic duct by a duodenoscope
  Other Names: Pancreatic duct stent (made of plastic material)
  Arms: Pancreatic stent

SUMMARY:
Dividing pancreas when performing left-sided resections opens the risk for leakage from the divided end of the pancreas. Pancreatic juices could have a severe effect on surrounding abdominal tissues with abscess formation producing systemic inflammation and potential lethal bleeding. Proper drainage of pancreatic juices is the primary treatment. Effective drainage reduces healing time. A pancreatic stent could theoretically improve the drainage of pancreatic juice into the duodenum and by this shorten the healing time still further.

Pre operative prophylactic stenting of the pancreas before division of the parenchyma has not shown a positive effect on fistula formation.

In an open randomized multicenter clinical trial we want to test the hypothesis that a reduced fistula healing time, in left sided pancreatic resections, could be reduced by introducing a pancreatic stent when on post operative day 3 or later a B och C fistula (according to the International Study Group on Pancreatic Fistula, ISGPF) is diagnosed by randomizing between pancreatic stent with drains versus only drains.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Left sided or distal pancreatic resection
* Grade B or C fistula on postoperative day 3 or later

Exclusion Criteria:

* Do not want to participate in study
* Can not read patient information in swedish
* The papilla can not be endoscopically reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
POPF healing time (days) | 12 days (median hospital stay)
  Post operative pancreatic fistula(POPF) and grade (A,B,C) is diagnosed according to ISGPF on post operative day 3 or later if the pancrease-amylase concentration is more than three times the upper limit of the normal plasma concentration of pancreas-amylase. When the drain fluid concentration is below this value the fistula is defined as healed.

SECONDARY OUTCOMES:
POPF grade (A,B,C) | 12 days (median hospital stay)
  International Study Group on Pancreatic Fistula (ISGPF) (Bassi et al 2005)defines fistula grade A-C. Grade A is leakage of pancreatic juice with a concentration of more than 3 times the upper normal level in plasma but no other clinical implication for the patient. If an inflammatory response is seen, but not sepsis, it is graded as B fistula and if sepsis occurs and/or single- or multi-organ dysfunction is seen it is graded as C.

OTHER OUTCOMES:
Blood chemistry | 12 days (median hospital stay)
  C-reactive protein, white blood cell count and pancreas amylase in plasma and drains
Morbidity | 12 days (median in hospital stay)
  Classification according to Clavien-Dindo
Mortality | < 90 days after the operation
Hospital stay | 12 days (median hospital stay)
  Number of days in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Dep of Surgical Gastroenterology, Karolinska University Hospital, Stockholm, Sweden